CLINICAL TRIAL: NCT07103941
Title: Effectiveness of Interocclusal Aligner (IOA) on Preventing Occlusal Changes in Patients Treated With a Mandibular Advancement Device (MAD): A Preliminary Study
Brief Title: IOA Preventing Occlusal Changes With MAD Use
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Isabel Moreno Hay (Other)
Collaborators: American Academy of Orofacial Pain (Unknown)
Responsible Party: Sponsor-Investigator, Isabel Moreno Hay, Associate Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 103755
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Sleep Related Breathing Disorder; Snoring; Obstructive Sleep Apnea (OSA); Open Bite; Occlusal Changes; Tooth Migration; Posterior Open Bite
Keywords: Interocclusal Aligner; Mandibular advancement Device; Posterior Open Bite; Occlusal Changes; Dental Changes; Protrusion; Sleep Appliance; Obstructive Sleep Apnea
MeSH Terms: conditions — Snoring; Sleep Apnea, Obstructive; Open Bite; Tooth Migration | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Parallel Assignment: Parallel Assignment Participants in this randomized clinical trial will be assigned to one of two parallel groups receiving standard-of-care interventions aimed at preventing occlusal changes during Mandibular Advancement Device (MAD) therapy for sleep-related breathing disorders. One group will use an interocclusal aligner (a morning repositioning device) after removing the MAD each morning. The other group will perform a daily set of jaw exercises designed to restore habitual occlusion.
  Each participant will remain in their assigned group for the duration of the 3-month study period, and no crossover between groups will occur. This parallel design allows for a direct comparison of the effectiveness of these two standard-of-care approaches in maintaining occlusal stability during MAD therapy.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Interocclusal Aligner (Active Comparator): Arm 1 (Interocclusal Aligner Group):
  "Morning Interocclusal Aligner to Maintain Occlusion" Participants in this arm will use a prefabricated thermoplastic device called the AM Aligner each morning immediately after removing their Mandibular Advancement Device (MAD). The aligner will be warmed and then gently bitten into for 2-5 minutes to help reposition the mandible and maintain the original occlusion. This approach is a standard-of-care method aimed at minimizing occlusal changes associated with MAD therapy.
  Interventions: Device: AM Aligner
- Daily Jaw Exercises (Active Comparator): Participants in this arm will be instructed to perform a standardized set of jaw exercises each morning after removing their MAD. The exercises include side-to-side jaw movements, backward pressure (such as the "thinker's pose"), and gentle simulated clenching.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Device: AM Aligner — Intervention Name: AM Aligner (Interocclusal Aligner) Type: Device Manufacturer: (AM Aligner; TAP Sleep Care, Texas, USA)
  Description:
  The AM Aligner is a prefabricated, commercially available thermoplastic appliance designed to help patients return their mandible to a normal resting position after nighttime use of a Mandibular Advancement Device (MAD). In this study, the aligner will be used each morning immediately after removing the MAD. The participant will bite into the warmed aligner for 2-5 minutes to promote realignment of the mandible and occlusion. This approach aims to minimize or prevent occlusal changes, including posterior open bite and anterior shift, associated with prolonged MAD therapy.
  This intervention is distinct from the alternative study arm, which uses a set of guided jaw exercises instead of a physical appliance to achieve the same goal.
  The AM Aligner used in this study is a standard-of-care option and is FDA-cleared for this use. It is not investigational.
  Arms: Interocclusal Aligner
Behavioral: Exercise — Participants in this arm will perform a standardized set of jaw exercises for 5 minutes each morning immediately after removing their Mandibular Advancement Device (MAD). The exercises are intended to assist in reestablishing the natural occlusal relationship following overnight mandibular advancement.
  This routine includes the following movements:
  Side-to-side jaw movements Backward pressure to the chin (similar to a "thinker's pose") Gentle simulated clenching
  The exercises are performed once daily and take approximately 2-3 minutes to complete. This approach represents a standard-of-care method for minimizing occlusal changes associated with MAD therapy.
  Arms: Daily Jaw Exercises

SUMMARY:
This study is evaluating two standard-of-care strategies used to prevent bite changes (occlusal changes) in patients treated with a Mandibular Advancement Device (MAD) for sleep-related breathing disorders such as obstructive sleep apnea (OSA). While MAD therapy is effective, it can lead to changes in how the teeth fit together, including the development of a posterior open bite.

Participants in this study will be randomly assigned to one of two standard-of-care approaches: using an interocclusal aligner each morning after removing the MAD, or performing daily jaw exercises. Both methods aim to reduce the risk of occlusal changes.

The study will follow participants over a 3-month period and includes dental evaluations, 3D oral scans, and short daily surveys. Findings from this research may help guide best practices for preserving occlusion during MAD therapy.

DETAILED DESCRIPTION:
Sleep-related breathing disorders (SRBD) are a group of disorders characterized by abnormal breathing during sleep, and common SRBD conditions encompass primary snoring and obstructive sleep apnea (OSA). Obstructive sleep apnea (OSA) is characterized by recurring episodes of partial or complete upper airway obstruction during sleep. This condition can result in daytime exhaustion, cognitive impairments, diminished quality of life, and elevated risks of cardiovascular and cerebrovascular illnesses, as well as increased mortality. OSA has also been linked to the development and progression of painful conditions such as temporomandibular disorders (TMD) and other orofacial pain conditions.

Currently, continuous positive airway pressure (CPAP) is recognized as the most effective treatment for OSA. However, patients' compliance with CPAP therapy is low, and it is oftentimes not tolerated. Therefore, almost two decades ago, the American Academy of Sleep Medicine approved the use of mandibular advancement devices (MADs) as an alternative treatment option. MADs work by mechanically advancing the mandible and maintaining it in a forward position, thereby decreasing airflow resistance and preventing collapse of the upper airway during sleep. MADs are also used for the cosmetic management of primary snoring.

Despite the promise of MADs in treating SRBD, one of the drawbacks to long-term use is the development of dental side effects. These include palatal tipping of the maxillary incisors, forward tilting of the mandibular incisors, minor mesial shifting of the mandibular molars, and posterior teeth losing contact or developing a posterior open occlusal relationship (POOR). The development of a POOR secondary to MAD use has been estimated to affect approximately 10-12% of individuals using these devices. However, beyond investigating the prevalence of POOR, the long-term consequences remain largely unexplored, with limited studies available. It has been hypothesized that POOR can cause sustained shortening of the lateral pterygoid muscles. As a result, when the patient attempts to achieve maximum intercuspation, the front teeth make contact while the back teeth fail to do so, which can significantly hinder a patient's ability to chew properly, resulting in impaired masticatory function. While this phenomenon is often temporary, resolving within hours or days, in rare instances, it may become irreversible.

Traditionally, simple jaw exercises aiming to stretch the lateral pterygoid muscle are recommended to alleviate or correct these side-effects of MADs. However, an emerging clinical trend is the use of an interocclusal aligner (IOA) following the removal of the MAD to minimize dental side effects, rather than relying solely on jaw exercises. However, the effectiveness of IOAs to prevent the development of POOR secondary to the MAD has not yet been empirically demonstrated.

The interocclusal appliances (interocclusal aligner (IOA)) include a variety of personalized appliances and pre-manufactured devices designed to restore the mandible to its usual pre-treatment position. These tools function by re-calibrating the patient's bite into maximum intercuspation, guiding each tooth back into its original position. Additionally, biting pressure is applied to reposition the condyles, with the goal of re-establishing or preserving proper occlusal alignment in the morning after each night of MAD therapy. The guide is customized to fit the patient's maxillary and mandibular teeth in their pre-treatment maximum intercuspation. Moreover, these devices assist in reversing tooth position changes by providing additional exercises that stretch and engage the jaw muscles.

The interocclusal aligner (IOA) is prepared either chairside or in a laboratory before the patient begins using the oral appliance. These aligners can be fabricated using hard or soft materials, with processed acrylics or thermoplastics being the most commonly used. After wearing the sleep appliance overnight, patients are instructed to bite into the aligner each morning until proper alignment between the maxillary and mandibular teeth is achieved, for as long as necessary for the occlusion to normalize.

To the best of our knowledge, there is currently no scientific evidence to support the use of interocclusal aligner (IOA) to prevent the development of POOR secondary to MAD use. Establishing the efficacy of the interocclusal aligner (IOA) would require a future efficacy trial where patients receiving MAD are randomly assigned to receive either stretching exercises (the standard of care) or use of an interocclusal aligner (IOA). Yet, there are logistical and technological burdens that undermine the feasibility of running such a trial. These include questions regarding the ability to recruit and retain sufficient patients, and questions regarding the ability to accurately measure POOR outcomes (i.e., the primary outcome of interest).

Currently, the presence of POOR is usually assessed using 12-µm shim stock foil (Artus Corp., Englewood, NJ, USA). However, this method may be subjective and does not quantify or visualize the occlusal changes or teeth movements. With the implementation of a digital workflow in dentistry, intraoral scanners are now being utilized to obtain precise 3-dimensional (3D) records of the patient's arch dimensions and occlusion. Intraoral scanners can also produce heat map analysis of the occlusal changes that a patient undergoes as a result of the use of a mandibular device for the management of SRBD, but the use of intraoral heat maps to assess POOR outcomes following treatment with MADs has never yet been validated to our knowledge.

The proposed study aims to collect preliminary data to inform the feasibility and design of a future full-scale efficacy trial comparing the use of daily jaw stretching exercises versus an interocclusal aligner (AM Aligner, Airway Management, LLC) in preventing the development of a posterior open occlusal relationship (POOR) in patients undergoing treatment with mandibular advancement devices (MADs).

The specific aims of the current study are as follows:

* Aim 1: To determine the recruitment and retention rates of participants willing to enroll in a randomized clinical trial comparing stretching exercises to the use of an interocclusal aligner (IOA).
* Aim 2: To evaluate the reliability of intraoral scanning (IOS) in detecting and tracking occlusal changes, such as posterior open occlusal relationship, palatal tipping of the maxillary incisors, proclination of the mandibular incisors, and mesial shifting of the mandibular molars, by comparing positional dental changes to baseline 3D records.

In summary, mandibular advancement devices (MADs) are a promising treatment for SRBDs. However, the devices are associated with significant and impactful postural and occlusal oral remodeling side effects. Currently, there are no established methods to effectively treat these complications. Specifically, this research will explore the efficacy of morning occlusal guides in mitigating POOR, thereby improving the long-term outcomes and patient tolerance of MAD therapy.

ELIGIBILITY:
Inclusion Criteria:

* adult participants (≥18 years)
* diagnosed with SRBD and prescribed Mandibular Advancement Device (MAD) therapy
* Participants will include patients with well restored natural dentition with all posterior teeth, excluding third molars, one missing premolar secondary to orthodontic treatment.

Exclusion Criteria:

* pervious orthognathic surgery
* anterior cross bite
* posterior cross bite
* existing open bite or implant supported restorations
* tooth mobility
* significant dental caries or periodontitis
* severe bruxism
* planned upcoming dental work including caps, crowns, implants, or braces
* inadequate mandibular protrusion
* severe micrognathia
* large tori
* significant claustrophobia
* significant nasal obstruction
* large oropharyngeal masses or large tonsils

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11-17 (Actual); Primary Completion 2026-03-28 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants enrolled in the study | 3 months
  Recruitment will be measured by tracking the number of participants who agree to enroll in a randomized clinical trial comparing stretching exercises to the use of an interocclusal aligner (IOA).

SECONDARY OUTCOMES:
Change in posterior occlusal contact relationship from baseline | Baseline, 4 weeks from baseline, 12 weeks from baseline
  Intraoral scanning (IOS) and clinical occlusal assessment (using shim stock and articulating paper) will be used to detect the development of a posterior open occlusal relationship. Positional changes observed on follow-up scans will be compared to baseline 3D records and clinical measurements.
  Unit of Measure: Binary outcome (presence or absence of occlusal contact)

OTHER OUTCOMES:
Change in axial inclination of maxillary incisors from baseline | Baseline, 4 weeks from baseline, 12 weeks from baseline
  Palatal tipping of the maxillary incisors will be evaluated using IOS and confirmed by clinical examination. Changes in tooth angulation will be compared to baseline 3D scans and clinical records.
  Unit of Measure: Degrees of axial inclination
Change in axial inclination of mandibular incisors from baseline | Baseline, 4 weeks from baseline, 12 weeks from baseline
  Proclination of mandibular incisors will be assessed by comparing IOS findings to baseline 3D records and corresponding clinical measurements. Unit of Measure: Degrees of axial inclination
Change in Mesial shifting of mandibular molars from baseline | Baseline, weeks from baseline, 12 weeks from baseline
  Mesial displacement of mandibular molars will be measured using IOS and verified through clinical tooth position assessment, with comparisons made to baseline digital and clinical records.
  Unit of Measure: Millimeters (mm) of linear positional change

CONTACTS AND LOCATIONS:
Overall Officials: Isable Moreno Hay, MS, PhD, Study Director — University of Kentucky
Locations (1):
- Orofacial Pain Center - University of Kentucky - Kentucky Clinic, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No